CLINICAL TRIAL: NCT01106391
Title: A Multicenter, Open Label, Prospective, Non-Randomized Study Of INCRAFT™ In Subjects With Abdominal Aortic Aneurysms
Brief Title: A Multicenter, Open Label, Prospective, Non-Randomized Study Of INCRAFT™ In Subjects With AAA (INNOVATION)
Acronym: INNOVATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EE09-01
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2022-04

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Abdominal aortic aneurysm; AAA; Safety; Performance; Stent graft system; First in Human; Endovascular repair
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AAA stent graft system (Experimental): Cordis AAA stent graft system "INCRAFT TM"
  Interventions: Device: Cordis AAA stent graft system "INCRAFT TM"

INTERVENTIONS:
Device: Cordis AAA stent graft system "INCRAFT TM"

SUMMARY:
This study is a multi-center prospective, open label, non-randomized investigation of INCRAFT™ in subjects with abdominal aortic aneurysms.

The study will enroll up to 60 subjects in up to 7 sites in Germany and Italy.

DETAILED DESCRIPTION:
This study is a multi-center prospective, open label, non-randomized investigation of INCRAFT™ in subjects with abdominal aortic aneurysms. The study will enroll up to 60 subjects at 7 sites in Germany and Italy. All treated subjects will be evaluated at 1 month, 3 months (if applicable), 6 and 12 months, and annually for a total of 5 years post-procedure. An interim analysis will be conducted after the 25th enrolled subject reaches the 30-day follow up visit

ELIGIBILITY:
INCLUSION CRITERIA:

1. Subject is a male or infertile female > 18 years of age
2. Subject understands study requirements and treatment procedures and agrees to sign an informed consent form prior to any study procedures.
3. Subject is considered an appropriate candidate for open surgical repair of an abdominal aortic aneurysm.
4. Subject has at least one of the following:

   1. Abdominal aortic aneurysm ≥4.5 cm in women or ≥ 5 cm in men in diameter
   2. Aneurysm, which is >4 cm and which has increased in size by 0.5 cm within 6 months
   3. The maximum aortic diameter is ≥1.5 times that of the reference aortic diameter
   4. Saccular aneurysm
5. Subject has access vessel size compatible with vascular access techniques and potential accessories used with delivery profile of 14Fr
6. Subject aortic aneurysm neck is ≥15 mm in length
7. Subject iliac landing zone≥10mm in length
8. Subject has distal iliac landing sites with diameter ranges of 9-18mm
9. Subject proximal aortic attachment is between 20-27 mm in diameter.
10. Subject has a minimum overall AAA treatment length (from lowest renal artery to distal landing zone) of 140 mm.
11. Subject is willing to comply with all specified follow-up evaluations.

EXCLUSION CRITERIA:

1. Subject has one of the following:

   1. a dissecting or inflammatory aneurysm
   2. acutely ruptured aneurysm
   3. pararenal or leaking aneurysm
2. The supra-renal aorta at 2cm above the lowest renal aorta is not more than the nominal diameter of the aortic bifurcate prosthesis
3. Aortic length (lowest renal artery origin to the aortic bifurcation) of <8.7 cm
4. Circumferential thrombosis and/or calcification ≥50% in the aortic and iliac landing zones
5. Circumferential thrombosis and/or calcification ≥50% in the supra-renal aorta
6. Subject has aneurysm neck angulations that are >60° in the supra-renal and/or infra-renal locations
7. Aortic bifurcation ≤18mm in diameter
8. Acute vascular injury due to trauma
9. Subject has a known allergy to contrast medium
10. Subject has known allergy to nitinol, PET or PTFE
11. Subject has a need for emergent surgery
12. Subject has a contraindication to undergoing angiography
13. Subject has a thoracic aortic aneurysm that requires treatment
14. Subject has Infra-renal aortic dissection
15. Subject has an Iliac anatomy which would require occlusion of both internal iliac arteries
16. Subject has congenital abnormalities in which the placement of the stent-graft will cause occlusion of major arterial flow. Such abnormalities should be evaluated (e.g. angiography or CT) prior to treatment
17. Subject has unstable angina as defined by Braunwald angina classification
18. Subject has morbid obesity (BMI of >40.0) or other clinical conditions that severely inhibit visualization of the aorta
19. Subject has connective tissue disease (e.g., Marfan's or Ehler's-Danos syndrome)
20. Subject has known bleeding or hypercoagulable disorder
21. Subject has contraindication for anticoagulation
22. Subject with Stroke or MI or intracranial bleeding within 3 months prior to the procedure
23. Subject with renal insufficiency (creatinine > 2.0 mg/dl)
24. Subject has known or suspected active infection at the time of the index procedure (for ex. Pneumonia, acute virus infection, contaminated wounds etc)
25. Subject is currently taking systemic immunosuppressant therapy
26. Subject had a major surgical procedure within 30 days prior to procedure or planned within 30 days post procedure
27. Subject has a life expectancy less than 2 years
28. Subject is currently participating in another research study involving an investigational device or new drug
29. Other medical, social, or psychological issues that in the opinion of the investigator preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment
30. Subject with an existing AAA surgical graft and/or a AAA stent-graft system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, PhD, MD., Principal Investigator — Universität Leipzig - Herzzentrum
Locations (1):
- Universitat Leipzig Herzzentrum, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scheinert D, Pratesi C, Chiesa R, Coppi G, Brunkwall JS, Klarenbeek G, Cebrian A, Torsello G. First-in-human study of the INCRAFT endograft in patients with infrarenal abdominal aortic aneurysms in the INNOVATION trial. J Vasc Surg. 2013 Apr;57(4):906-14. doi: 10.1016/j.jvs.2012.09.079. Epub 2013 Jan 18. PMID 23332982
- [Background] Torsello G, Brunkwall J, Scheinert D. Cordis INCRAFT ultra-low profile AAA stent-graft system. J Cardiovasc Surg (Torino). 2011 Oct;52(5):661-7. PMID 21894137
- [Background] Coppi G, Njila M, Coppi G, Saitta G, Silingardi R, Pratesi C, Chiesa R, Scheinert D, Brunkwall JS, Torsello G. INCRAFT(R) Stent-Graft System: one-year outcome of the INNOVATION Trial. J Cardiovasc Surg (Torino). 2014 Feb;55(1):51-9. PMID 24356046
- [Background] Torsello G, Scheinert D, Brunkwall JS, Chiesa R, Coppi G, Pratesi C. Safety and effectiveness of the INCRAFT AAA Stent Graft for endovascular repair of abdominal aortic aneurysms. J Vasc Surg. 2015 Jan;61(1):1-8. doi: 10.1016/j.jvs.2014.06.007. Epub 2014 Jul 19. PMID 25053535
- [Derived] Torsello G, Pratesi G, van der Meulen S, Ouriel K; INNOVATION trial collaborators. Aortoiliac remodeling and 5-year outcome of an ultralow-profile endograft. J Vasc Surg. 2019 Jun;69(6):1747-1757. doi: 10.1016/j.jvs.2018.09.059. Epub 2018 Dec 24. PMID 30591290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 60 subjects enrolled in this trial at 7 sites in Germany and Italy from March 19, 2010 to June 20, 2011.
Pre-assignment Details: Of the 78 subjects consented and assessed for eligibility, 18 subjects did not meet all study entrance criteria and were considered screen failure.
Groups:
- The INCRAFT™ AAA Stent-graft System: The Cordis INCRAFT™ AAA stent-graft system is a modular bifurcated endovascular graft system that is used for the treatment of infrarenal abdominal aortic aneurysms (AAA). The system is constructed with self-expanding, nickel-titanium (nitinol) alloy stent rings and woven polyester graft tubes. The bifurcated aortic prosthesis includes a transrenal stent with integrated fixation barbs. The limbs include annular fabric crimps between the supporting stents.
Period: Overall Study
Arm/Group | The INCRAFT™ AAA Stent-graft System
Started | 60
Completed (Completed is defined as subjects completed 5 years follow up.) | 41
Not Completed | 19
Not completed — Death | 12
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (6.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 57
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 31
  Italy | 29
Body mass index [Mean (Standard Deviation); unit: kg/m²] | 26.7 (3.05)
Diabetes [Count of Participants; unit: Participants]
  Insulin-dependent diabetes | 3
  Non-insulin-dependent diabetes | 10
  Free of diabetes | 47
Hypertension [Count of Participants; unit: Participants]
  Hypertension | 57
  Free of Hypertension | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Technical Success Through the One Month Follow up.
Description: Technical success is defined as the successful deployment of the stent-graft to the desired location in the absence of Types I, III or IV endoleaks at the conclusion of the procedure and through the one month follow up.
Time Frame: From procedure to one month follow up
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 60
Participants | 54
Statistical Analysis 1: Comparison: The INCRAFT™ AAA Stent-graft System; Since this was a feasibility study without comparisons, sample size was not determined based on statistical consideration. No formal hypothesis testing was performed either; Test type: Superiority or Other; Rate of technical success (%) = 90, 95% CI 2-sided [79.5 to 96.2] — The 95% confidence interval was based on the exact confidence interval (Collett, 1991)

2. Primary Outcome: Rate of Primary Safety Endpoint Within 1 Month Post-procedure.
Description: Primary safety is defined by the absence of Types I, III or IV endoleaks and device and/or procedural related major adverse events within 1 month post-procedure. Major adverse events include death, MI, stroke and renal failure.
Time Frame: One month follow-up
Population: The analysis population consists of subjects with complete core laboratory data at 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 58
Participants | 56
Statistical Analysis 1: Comparison: The INCRAFT™ AAA Stent-graft System; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate of achieved primary safety(%) = 97, 95% CI 2-sided [88.1 to 99.6] — The 95% confidence interval was based on the exact confidence interval (Collett, 1991)

3. Secondary Outcome: Percentage of Participants With Incidence of Aneurysm Enlargement Annually Through 5 Years Post - Procedure.
Description: Incidence of aneurysm enlargement annually through 5 years post - procedure. Aneurysm enlargement is defined as being compared to the 30 day baseline assessment.
Time Frame: Day 30 through year 5 post-procedure
Population: All enrolled subjects. However at each annual assessment of aneurysm enlargement, the numbers of follow-up subjects are 53, 50, 45, 39, 38 at year 1 through 5 respectively.
Measure: Number; unit: percentage of subjects with endpoint
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 60
percentage of subjects with endpoint
  Year 1: number analyzed (Participants) | 53
  Year 1 | 0.0
  Year 2: number analyzed (Participants) | 50
  Year 2 | 0.0
  Year 3: number analyzed (Participants) | 45
  Year 3 | 4.4
  Year 4: number analyzed (Participants) | 39
  Year 4 | 10.3
  Year 5: number analyzed (Participants) | 38
  Year 5 | 7.9

4. Secondary Outcome: Percentage of Participants With Incidence of Stent-graft Migration Annually Through 5 Years Post - Procedure.
Description: Incidence of Stent-graft Migration annually through 5 years post - procedure. Stent-graft Migration is defined as being compared to the 30 day baseline assessment.
Time Frame: Day 30 through year 5 post-procedure
Population: All enrolled subjects. However at each annual assessment of Stent-graft Migration, the numbers of follow-up subjects are 53, 50, 44, 38, 37 at year 1 through 5 respectively.
Measure: Number; unit: percentage of subjects with endpoint
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 60
percentage of subjects with endpoint
  Year 1: number analyzed (Participants) | 53
  Year 1 | 0.0
  Year 2: number analyzed (Participants) | 50
  Year 2 | 0.0
  Year 3: number analyzed (Participants) | 44
  Year 3 | 0.0
  Year 4: number analyzed (Participants) | 38
  Year 4 | 0.0
  Year 5: number analyzed (Participants) | 37
  Year 5 | 0.0

5. Secondary Outcome: The Cumulative Percentage of Participants With Major Adverse Events at Annually Through 5 Years Post - Procedure.
Description: The cumulative percentage of participants with Major Adverse Events (MAE) at annually through 5 years post - procedure; i.e., the percentage of MAE at Year 1 includes all MAEs occurred during the first year, the percentage at Year 2 includes all MAEs during the first two years, and etc. The Major adverse events include death, stroke, Q wave myocardial infarction, and renal failure
Time Frame: From day 1 through year 5 post-procedure
Population: All enrolled subjects. However at each annual assessment of major adverse events, the numbers of follow-up subjects are 56, 52, 55, 51 and 50 at year 1 through 5 respectively.
Measure: Number; unit: The cumulative percentage of Participant
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 60
The cumulative percentage of Participant
  Year 1: number analyzed (Participants) | 56
  Year 1 | 1.8
  Year 2: number analyzed (Participants) | 52
  Year 2 | 11.5
  Year 3: number analyzed (Participants) | 55
  Year 3 | 12.7
  Year 4: number analyzed (Participants) | 51
  Year 4 | 17.6
  Year 5: number analyzed (Participants) | 50
  Year 5 | 24

6. Secondary Outcome: The Percentage of Participants With Endoleaks at Annually Through 5 Years Post - Procedure.
Description: The percentage of endoleaks at annually through 5 years post - procedure. Endoleak contains Types I and III endoleaks
Time Frame: From day 1 through year 5 post-procedure
Population: All enrolled subjects. However at each annual assessment of endoleaks, the numbers of follow-up subjects are 53, 50, 45, 39, 38 at year 1 through 5 respectively.
Measure: Number; unit: percentage of subjects with endpoint
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 60
percentage of subjects with endpoint
  Year 1: number analyzed (Participants) | 53
  Year 1 | 0.0
  Year 2: number analyzed (Participants) | 50
  Year 2 | 0.0
  Year 3: number analyzed (Participants) | 45
  Year 3 | 4.4
  Year 4: number analyzed (Participants) | 39
  Year 4 | 2.6
  Year 5: number analyzed (Participants) | 38
  Year 5 | 2.6

7. Secondary Outcome: The Percentage of Participants With Stent-graft Fractures at 30 Days and Annually Through 5 Years Post - Procedure.
Description: The percentage of stent-graft fracture at 30 days and annually through 5 years post - procedure. Stent-graft fracture is defined as stent skeleton fracture and barb separation
Time Frame: From day 1 through year 5 post-procedure
Population: All enrolled subjects. However at each assessment of stent-graft fracture , the numbers of follow-up subjects are 54, 52, 46, 43, 40, 39 at 30 days and at year 1 through 5 respectively.
Measure: Number; unit: percentage of subjects with endpoint
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 60
percentage of subjects with endpoint
  Day 30: number analyzed (Participants) | 54
  Day 30 | 0.0
  Year 1: number analyzed (Participants) | 52
  Year 1 | 0.0
  Year 2: number analyzed (Participants) | 46
  Year 2 | 0.0
  Year 3: number analyzed (Participants) | 43
  Year 3 | 1.0
  Year 4: number analyzed (Participants) | 40
  Year 4 | 2.5
  Year 5: number analyzed (Participants) | 39
  Year 5 | 2.6

8. Secondary Outcome: The Percentage of Participants With Thrombosis at 30 Days and Annually Through 5 Years Post - Procedure.
Description: The percentage of Thrombosis at hospital discharge at 30 days and annually through 5 years post - procedure.
Time Frame: From day 1 through year 5 post-procedure
Population: All enrolled subjects. However at each assessment of thrombosis , the numbers of follow-up subjects are 58, 56, 52, 55, 51, 50 at 30 days and at year 1 through 5 respectively.
Measure: Number; unit: percentage of subjects with endpoint
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 60
percentage of subjects with endpoint
  Day 30: number analyzed (Participants) | 58
  Day 30 | 0.0
  Year 1: number analyzed (Participants) | 56
  Year 1 | 0.0
  Year 2: number analyzed (Participants) | 52
  Year 2 | 1.9
  Year 3: number analyzed (Participants) | 55
  Year 3 | 1.8
  Year 4: number analyzed (Participants) | 51
  Year 4 | 2.0
  Year 5: number analyzed (Participants) | 50
  Year 5 | 2.0

9. Secondary Outcome: The Percentage of Participants With Stent Graft Explant at 30 Days and Annually Through 5 Years Post - Procedure.
Description: The percentage of Stent Graft Explant at hospital discharge at 30 days and annually through 5 years post - procedure.
Time Frame: From day 1 through year 5 post-procedure
Population: All enrolled subjects. However at each assessment of thrombosis , the numbers of follow-up subjects are 58, 55, 52, 55, 51, 50 at 30 days and at year 1 through 5 respectively.
Measure: Number; unit: percentage of subjects with endpoint
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 60
percentage of subjects with endpoint
  Day 30: number analyzed (Participants) | 58
  Day 30 | 0.0
  Year 1: number analyzed (Participants) | 55
  Year 1 | 0.0
  Year 2: number analyzed (Participants) | 52
  Year 2 | 0.0
  Year 3: number analyzed (Participants) | 55
  Year 3 | 0.0
  Year 4: number analyzed (Participants) | 51
  Year 4 | 0.0
  Year 5: number analyzed (Participants) | 50
  Year 5 | 0.0

10. Secondary Outcome: The Percentage of Participants With Endoleg Patency at 30 Days and Annually Through 5 Years Post - Procedure.
Description: The percentage of participants with Endoleg Patency by CT scan at 30 days and annually through 5 years post - procedure.
Time Frame: From day 1 through year 5 post-procedure
Population: All enrolled subjects. However at each assessment of stent-graft fracture , the numbers of follow-up subjects are 58, 53, 45, 45, 41, 39 at 30 days and at year 1 through 5 respectively.
Measure: Number; unit: percentage of subjects with endpoint
Arm/Group | The INCRAFT™ AAA Stent-graft System
Number analyzed (Participants) | 60
percentage of subjects with endpoint
  Day 30: number analyzed (Participants) | 58
  Day 30 | 100
  Year 1: number analyzed (Participants) | 53
  Year 1 | 100
  Year 2: number analyzed (Participants) | 45
  Year 2 | 100
  Year 3: number analyzed (Participants) | 45
  Year 3 | 97.8
  Year 4: number analyzed (Participants) | 41
  Year 4 | 97.6
  Year 5: number analyzed (Participants) | 39
  Year 5 | 97.4

ADVERSE EVENTS:
Time Frame: From Day 1 through 5 years post-procedure
Arm/Group | The INCRAFT™ AAA Stent-graft System
Serious Adverse Events (participants affected / at risk) | 8/60
Other Adverse Events (participants affected / at risk) | 44/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The INCRAFT™ AAA Stent-graft System (N=60)
Hematoma / bleeding puncture site - major (Injury, poisoning and procedural complications) | 2 (2)
Pleural effusion (Infections and infestations) | 1 (1)
strong lymphatic wound secretions without infection (Blood and lymphatic system disorders) | 1 (1)
Claudication (Vascular disorders) | 1 (1)
Dissection (Vascular disorders) | 1 (1)
Lymphocele right groin postoperatively (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Myocardial infarction (Vascular disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The INCRAFT™ AAA Stent-graft System (N=60)
Hematoma/bleeding puncture site - minor (Injury, poisoning and procedural complications) | 1 (1)
Pseudo aneurysm (Injury, poisoning and procedural complications) | 1 (1)
Arrhythmia - Bradycardia (Cardiac disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Prosthesis leaks (endoleak I) (General disorders) | 1 (1)
Prosthesis leaks (endoleak IV) (General disorders) | 4 (4)
Prosthesis occlusion/ stenosis (Vascular disorders) | 1 (1)
Atherosclerosis (Vascular disorders) | 1 (1)
Perforation (Vascular disorders) | 1 (1)
Fever (General disorders) | 24 (24)
Hematuria (Renal and urinary disorders) | 1 (1)
Post-implant syndrome (General disorders) | 3 (3)
Arterial occlusion (Vascular disorders) | 2 (2)
Hematoma/bleeding (Injury, poisoning and procedural complications) | 1 (1)
Fever (General disorders) | 1 (1)
High creatinine level (Investigations) | 1 (1)
Endoleak, type undetermined (General disorders) | 1 (1)
Asymptomatic lymphocele (Blood and lymphatic system disorders) | 1 (1)
Stent misplacement (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Small infarct right kidney (Renal and urinary disorders) | 1 (1)
Periprocedural red cells transfusion (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days